CLINICAL TRIAL: NCT02168855
Title: Cessation in Non-Daily Smokers: A RCT of NRT With Ecological Momentary Assessment
Brief Title: Cessation in Non-Daily Smokers
Acronym: QUITS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brian Primack (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Brian Primack, MD, PhD, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1R01DA034629 (NIH)
Record Dates: First submitted 2014-06-18; First posted 2014-06-20 (Estimated); Results first posted 2020-05-06 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-04

CONDITIONS: Smoking
Keywords: Smoking cessation; Non-daily smokers; Ecological Momentary Assessment; nicotine replacement therapy
MeSH Terms: conditions — Smoking; Smoking Cessation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active nicotine gum (Active Comparator)
  Interventions: Drug: active nicotine gum; Behavioral: Standard behavioral therapy
- Inactive gum (Placebo Comparator)
  Interventions: Behavioral: Standard behavioral therapy

INTERVENTIONS:
Drug: active nicotine gum — 2 mg, standard over-the-counter nicotine replacement therapy gum
  Arms: Active nicotine gum
Behavioral: Standard behavioral therapy — Standard behavioral therapy for smoking cessation

SUMMARY:
The purpose of this study is to examine the effect of as-needed oral Nicotine Replacement Therapy (NRT) - 2 mg nicotine gum - for smoking cessation in non-daily, or intermittent, smokers, and to study the process of relapse in ITS, using Ecological Momentary Assessment (EMA).

DETAILED DESCRIPTION:
Our aim is to study the effect of as-needed oral Nicotine Replacement Therapy (NRT) - 2 mg nicotine gum - for smoking cessation in non-daily, or intermittent, smokers (ITS), and to study the process of relapse in ITS, using Ecological Momentary Assessment (EMA). This is a double-blind, randomized, placebo-controlled trial of oral NRT for smoking cessation in ITS. 600 ITS who are interested in quitting will be recruited through multiple channels. Enrollees will be randomized 1:1 to active 2 mg nicotine gum or an inert control gum. Participants will attend 6 sessions with brief behavioral support, with a planned quit day at week 2. Short and long term abstinence will be assessed and biochemically validated. EMA data collection includes two weeks of baseline data on ad lib smoking patterns and 6 weeks of post-quit data. This will capture data on craving, withdrawal, and relapse among ITS, and relate relapse contexts to baseline smoking patterns.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Smoking for at least 3 years
* Smoking non-daily for at least one year (< or = 27 days/month)
* Smoke at least weekly
* Intention to quit smoking within the next month and a desire to receive behavioral and medication treatment
* Willing and able to come to the laboratory for 8 visits over a 14-week period, as well as a ninth and final visit 6 months after their quit date
* Willing to monitor behavior via an electronic diary for 8 weeks
* Able to read and write English (in order to understand questionnaires and study instructions)

Exclusion Criteria:

* Regular use of any form of tobacco other than cigarettes
* Recent or severe mental illness (uncontrolled severe depression or mood symptoms, active hallucinations, and or hospitalization in the past month for a psychiatric condition)
* Night and/or 'swing' shift work (which complicates EMA schedules)
* Known plans to relocate or move from the Pittsburgh area within the coming 6 months
* Received cessation treatment within past year
* Use of bupropion or varenicline in past 2 months
* Past use of nicotine gum (to avoid un-blinding)
* Contraindication to NRT
* (for women) Current pregnancy or breastfeeding or plan to become pregnant during the next 2 months
* Member of the same household already participating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 505 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian A Primack, MD, PhD, Principal Investigator — University of Pittsburgh, Division of General Internal Medicine
Locations (1):
- Smoking Research Group, University of Pittsburgh, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: While 505 participants were enrolled in and began the study, only 369 of these were ultimately randomized to the active nicotine gum or inactive (placebo) gum arms. Those who were not randomized due to either participant-initiated drop out (n=36), research-team-initiated withdrawal due to noncompliance (n=83), or loss to followup (n=17).
Period: Overall Study
Arm/Group | Active Nicotine Gum | Inactive Gum
Started | 181 | 188
Completed | 169 | 177
Not Completed | 12 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Nicotine Gum | Inactive Gum | Total
Number analyzed (Participants) | 181 | 188 | 369
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.72 (13.76) | 45.87 (15.02) | 44.32 (14.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108 | 102 | 210
  Male | 73 | 86 | 159
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 9 | 20
  Not Hispanic or Latino | 170 | 179 | 349
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 6 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 67 | 81 | 148
  White | 94 | 93 | 187
  More than one race | 11 | 8 | 19
  Unknown or Not Reported | 3 | 3 | 6
Cigarettes smoked per day on average, assessed over the last 28 days, including all days [Mean (Standard Deviation); unit: cigarettes per day] — Collected via self-reported "time-line follow-back" calendar, in which participants reported on each day in the previous 28 days the number of cigarettes they smoked. The average is calculated as the number of cigarettes smoked per days, including each day of the previous 28 days in the denominator, regardless of whether the participant reported smoking on each of those days. In other words, if a participant reported smoking on only 4 of the past 28 days, the average would be calculated by adding the total number of cigarettes smoked on those 4 days and dividing that number by 28.
  cigarettes per day | 1.8 (1.5) | 1.9 (1.5) | 1.9 (1.5)
Cigarettes smoked per day on average, assessed over the last 28 days, including only smoking days [Mean (Standard Deviation); unit: cigarettes per day] — Collected via self-reported "time-line follow-back" calendar, in which participants reported on each day in the previous 28 days the number of cigarettes they smoked. The average is then calculated, to arrive at this measure - the number of cigarettes smoked per day, at baseline, including in the denominator only the number of days the participant reported having smoked. In other words, if a participant reported smoking on only 4 of the past 28 days, the average would be calculated by adding the total number of cigarettes smoked on those 4 days, and dividing that number by 4.
  cigarettes per day | 3.3 (2.0) | 3.9 (2.9) | 3.6 (2.5)

OUTCOME MEASURES:

1. Primary Outcome: Smoking Cessation, Continuous 6-month Abstinence
Description: Long term abstinence assessed and biochemically validated. The results reported are the number of participants self-reporting continuous abstinence throughout the 6-month, post-quit follow-up period. To be considered abstinent, a participant must have self-reported having not smoked during this period, demonstrated carbon monoxide levels less than or equal to 3 at each study visit, and cotinine values assessed via urinalysis at levels less than or equal to 25 ng/ml.
Time Frame: up to week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Active Nicotine Gum | Inactive Gum
Number analyzed (Participants) | 181 | 188
Participants | 13 | 10
Statistical Analysis 1: Comparison: Active Nicotine Gum vs Inactive Gum; Test type: Superiority; p = 0.46, Regression, Logistic; This is a logistic regression model of the active versus placebo arm, while controlling for age and cigarettes smoked per day at enrollment; Odds Ratio (OR) = 1.39, 95% CI 2-sided [0.58 to 3.29] — The active arm is the numerator and the placebo arm is the denominator of the odds ratio

2. Secondary Outcome: Characteristics of Quit and Relapse Process - Craving
Description: Ecological Momentary Assessment (EMA) methods will be used to study the craving, withdrawal, and relapse processes among ITS and relate relapse contexts to baseline smoking patterns. This measure assessed the intensity of craving experienced by participants during their attempt to quit smoking, via self-report. To ensure the results were not influenced by the use of active nicotine replacement gum, only the participants receiving inactive gum (containing no nicotine) are included in this analysis.
  The scale's range was 0-100, with higher values reflecting higher levels of self-reported craving (maximum score of 100), whereas a score of 0 indicates no craving. "Background" craving is defined as that experienced when a participant was not smoking or feeling a temptation to smoke. "Temptations to smoke" refers to situations where a participant was tempted to smoke and did, or tempted to and did not.
Time Frame: Six-week post-quit period
Population: This is the subset of placebo arm ITS participants who had achieved initial abstinence. These participants all submitted at least one background and one temptation report. To ensure the results were not influenced by using active nicotine gum, only participants receiving inactive gum (containing no nicotine) are included in this analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Inactive Gum: Momentary real-time report of situational and mood and craving factors, randomly assessed throughout the day, at times not associated with smoking, use of other nicotine products, temptation to smoke, or use of gum
Arm/Group | Inactive Gum
Number analyzed (Participants) | 130
score on a scale
  Background | 16.68 (1.61)
  Temptations to smoke | 57.09 (2.50)
Statistical Analysis 1: Comparison: Inactive Gum; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Includes random subject intercept effect; Odds Ratio (OR) = 1.90, 95% CI 2-sided [1.83 to 1.98] — Reflects an odds ratio relative to a 10-unit increase in craving. Temptations are the numerator and background is the denominator

3. Secondary Outcome: Characteristics of Quit and Relapse Process - Negative Affect
Description: Ecological Momentary Assessment (EMA) methods will be used to study the craving, withdrawal, and relapse processes among ITS and relate relapse contexts to baseline smoking patterns. This measure assesses the intensity of negative affect participants experienced during their attempt to quit smoking. To ensure the results were not influenced by the use of active nicotine replacement gum, only the participants receiving inactive gum (containing no nicotine) are included in this analysis.
  The scale's range was 0-100, with higher values reflecting higher levels of self-reported negative affect (maximum score of 100), whereas a score of 0 would indicate no negative affect. 50 indicates the population mean with a standard deviation of 10. "Background" reports are defined as those experienced when a participant was not smoking or feeling a temptation to smoke. "Temptations to smoke" refers to situations where a participant was tempted to smoke and did, or tempted to and did not.
Time Frame: Six-week post-quit period
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Inactive Gum
Number analyzed (Participants) | 130
T-score
  Background | 49.13 (0.63)
  Temptations to smoke | 51.96 (0.84)
Statistical Analysis 1: Comparison: Inactive Gum; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Includes random subject intercept effect; Odds Ratio (OR) = 1.66, 95% CI 2-sided [1.51 to 1.83] — Reflects an odds ratio relative to a 10-unit increase in negative affect T-score. Temptations are the numerator and background is the denominator

4. Secondary Outcome: Characteristics of Quit and Relapse Process - Saw No Smoking Cues
Description: Ecological Momentary Assessment (EMA) methods will be used to study the craving, withdrawal, and relapse processes among ITS and relate relapse contexts to baseline smoking patterns.To ensure the results were not influenced by the use of active nicotine replacement gum, only the participants receiving inactive gum (containing no nicotine) are included in this analysis.
  This measure reports the percentage of instances during which participants were not exposed to physical cues to smoke, such as cigarettes, ashtrays, or lighters), when experiencing temptations to smoke compared to experiencing no temptations to smoke. "Background" reports are defined as those experienced when a participant was not smoking or feeling a temptation to smoke. "Temptations to smoke" refers to situations where a participant was tempted to smoke and did, or tempted to and did not.
Time Frame: Six-week post-quit period
Population: as for outcome 2
Measure: Number; unit: percentage of assessments
Groups:
- Background: Momentary real-time report of situational and mood and craving factors, randomly assessed throughout the day, at times not associated with smoking, use of other nicotine products, temptation to smoke, or use of gum
Arm/Group | Background
Number analyzed (Participants) | 130
percentage of assessments
  Background | 83.64
  Temptations to smoke | 59.11
Statistical Analysis 1: Comparison: Background; Test type: Superiority; p < 0.0001, Regression, Logistic; Includes random subject intercept effect; Odds Ratio (OR) = 0.18, 95% CI 2-sided [0.14 to 0.21] — Odds ratio where temptations are the numerator and background is the denominator, that no smoking cues were seen

5. Secondary Outcome: Characteristics of Quit and Relapse Process - No Others Smoking Nearby
Description: Ecological Momentary Assessment (EMA) methods will be used to study the craving, withdrawal, and relapse processes among ITS and relate relapse contexts to baseline smoking patterns. To ensure the results were not influenced by the use of active nicotine replacement gum, only the participants receiving inactive gum (containing no nicotine) are included in this analysis.
  This measure reports the percentage of instances during which participants were not exposed to others smoking nearby, when experiencing temptations to smoke compared to experiencing no temptations to smoke. "Background" reports are defined as those experienced when a participant was not smoking or feeling a temptation to smoke. "Temptations to smoke" refers to situations where a participant was tempted to smoke and did, or tempted to and did not.
Time Frame: Six-week post-quit period
Population: as for outcome 2
Measure: Number; unit: percentage of assessments
Arm/Group | Background
Number analyzed (Participants) | 130
percentage of assessments
  Background | 90.42
  Temptations to smoke | 66.82
Statistical Analysis 1: Comparison: Background; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 0.19, 95% CI 2-sided [0.15 to 0.23] — Odds ratio where temptations are the numerator and background is the denominator, that no other people were seen smoking nearby

ADVERSE EVENTS:
Time Frame: Data for adverse events was collected over the period of time during which each participant was enrolled and participating in the study. For participants completing the entire study, this period would be approximately 26 weeks - i.e., during the 2 weeks during which baseline data was collected, and the 24 weeks that began with their quit date and continued on for the following 6 months.
Description: Adverse events were assessed during study visits via in-session interactions in which study participants were prompted to describe their experiences since the prior visit in an open-ended format and answers were recorded by research assistants within study session tracking assessment forms.
Arm/Group | Active Nicotine Gum | Inactive Gum
All-Cause Mortality (participants affected / at risk) | 0/181 | 0/188
Serious Adverse Events (participants affected / at risk) | 9/181 | 14/188
Other Adverse Events (participants affected / at risk) | 93/181 | 65/188
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Nicotine Gum (N=181) | Inactive Gum (N=188)
Hospitalization for gastrointestinal viral infection (Gastrointestinal disorders) | 2 (2) | 0 (0)
Hospitalization for pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Foot surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Surgery for Appendicitis (Surgical and medical procedures) | 1 (1) | 0 (0)
Hemorrhoidectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Hospitalization for lupus flare-up (Immune system disorders) | 1 (1) | 0 (0)
Hospitalization for GERD flare-up (Gastrointestinal disorders) | 1 (1) | 0 (0)
Surgery on ovaries (Surgical and medical procedures) | 1 (1) | 0 (0)
Worsening of degenerative disc disease (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hospitalization for wrist injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Carpal tunnel surgery (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Root canal (Surgical and medical procedures) | 0 (0) | 1 (1)
Hospitalization for after car accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hospitalization for high blood pressure (Vascular disorders) | 0 (0) | 1 (1)
Worsening of lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Broken hip (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Breast cancer (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Hospitalization for allergic skin reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hospitalization for thyroid disorder (Endocrine disorders) | 0 (0) | 1 (1)
Corneal implant surgery (Eye disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Nicotine Gum (N=181) | Inactive Gum (N=188)
Gastric upset (Gastrointestinal disorders) | 28 (28) | 13 (13)
Weight gain (Metabolism and nutrition disorders) | 14 (14) | 15 (15)
Headache (General disorders) | 15 (15) | 13 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 14 (14)
Irritability (General disorders) | 13 (13) | 7 (7)
Throat or mouth irritation (General disorders) | 13 (13) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-01-08): https://cdn.clinicaltrials.gov/large-docs/55/NCT02168855/SAP_000.pdf
  • Study Protocol (2016-06-02): https://cdn.clinicaltrials.gov/large-docs/55/NCT02168855/Prot_001.pdf